CLINICAL TRIAL: NCT06744023
Title: The Effect of Improved Envıronment Accordıng to Watson's Theory of Human Care on Sleep, Anxıety, and Depressıon ın Patıents Undergoıng Open Heart Surgery: A Randomızed Controlled Study
Brief Title: Effects of Improved Environment on Sleep, Anxiety-Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hatice AZİZOĞLU (Other)
Responsible Party: Sponsor-Investigator, Hatice AZİZOĞLU, Assistant Professor, Yuzuncu Yil University
Organization: Yuzuncu Yil University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2023/09-17
Record Dates: First submitted 2024-06-20; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Coronary Disease; Cardiovascular Diseases
Keywords: Open heart surgery; anxiety; depression; improved environment; sleep quality; sleep duration
MeSH Terms: conditions — Coronary Disease; Cardiovascular Diseases; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial. Upon admission to the ward from the postoperative intensive care unit, the experimental group underwent environmental remediation for three days. The environmental arrangements ensured that the patient room maintained an appropriate temperature range of 18-26 °C and humidity values of 30-60%. Monitoring took place at 21:00, 22:00, and 23:00 on Days 1, 2, and 3. On Days 1, 2, and 3, the patient room's light brightness gradually decreased at 21:00, 22:00, and 23:00. On the morning of the fourth day, the patients were interviewed face-to-face, and the research questionnaires were filled out.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERIMENTAL GROUP (Experimental): Upon admission to the ward from the postoperative intensive care unit, the experimental group underwent environmental remediation for three days. The environmental arrangements ensured that the patient room maintained an appropriate temperature range of 18-26 °C and humidity values of 30-60%. Monitoring took place at 21:00, 22:00, and 23:00 on Days 1, 2, and 3. On Days 1, 2, and 3, the patient room's light brightness gradually decreased at 21:00, 22:00, and 23:00. On the morning of the fourth day, the patients were interviewed face-to-face, and the research questionnaires were filled out.
  Interventions: Other: To examine the effect of the improved environment according to Watsons Human Care Theory on sleep quality, anxiety, and depression in patients undergoing open heart surgery.
- CONTROL GROUP (No Intervention): The patients in the control group continued to receive standard treatment and care. On the morning of the fourth day after the patients were admitted to the ward from the postoperative intensive care unit, the patients were interviewed face-to-face and the Personal Information Form, RCSQ, and HAD Scale were completed.

INTERVENTIONS:
Other: To examine the effect of the improved environment according to Watsons Human Care Theory on sleep quality, anxiety, and depression in patients undergoing open heart surgery. — The patients who underwent open heart surgery and who were in the experimental group were admitted to the ward from the postoperative intensive care unit and the environment was improved for three days based on the improved environment of Watson's HCT, and on the morning of the fourth day in the clinic, the patients were interviewed face to face and the Personal Information Form, RSCQ and HAD Scale were completed. The following improvements were implemented within the scope of environmental improvement:
  * Considering the seasonal conditions, the patient room was ensured to have appropriate temperature (18-26 °C) and humidity values (30-60%), and the temperature and humidity were gradually reduced and maintained in the appropriate range by monitoring at 21:00, 22:00, and 23:00 (Days 1, 2, and 3)
  * In line with the environmental arrangements, the brightness of the light in the patient room was gradually reduced at 21:00, 22:00, and 23:00 using the Light Meter LM-3000 (Days 1, 2, and 3)
  Other Names: Improve environment
  Arms: EXPERIMENTAL GROUP

SUMMARY:
The aim of this randomized controlled trial was to examine the effect of an improved environment on sleep, anxiety, and depression in patients undergoing open heart surgery. This study aims to answer the following main questions:

* According to Watson's Human Care Theory, what is the effect of the improved environment on patients' sleep level and sleep quality?
* According to Watson's Human Care Theory, what is the effect of the improved environment on patients' anxiety and depression levels?

In order to observe the effect of the improved environment on sleep, anxiety, and depression, the researchers ensured that the room temperature, humidity, and lumen range of the light were at the appropriate level in the first 3 days after the surgery of the patients in the experimental group and gradually decreased them gradually.

DETAILED DESCRIPTION:
The aim of this randomized controlled trial was to examine the effect of an improved environment on sleep, anxiety, and depression in patients undergoing open heart surgery. This study aims to answer the following main questions:

* According to Watson's Human Care Theory, what is the effect of the improved environment on patients' sleep level and sleep quality?
* According to Watson's Human Care Theory, what is the effect of the improved environment on patients' anxiety and depression levels? Before collecting data for this study, the "G. Power-3.1.9.2" program calculated the sample size at an 80% confidence level. The "Sample Calculation Formula with Known Universe (Population Volume)" (n = Nz2pq / d2(N-1) + z2pq) determined the sample. The literature review determined the "effect size" value to be 0.096. Taking the primary type error of 5% (Z = 1,96), the test power of 80%, and the effect size value of 0,096 units, we calculated the minimum sample size as n = 60. Therefore, the study included 60 volunteer patients, with 30 placed in the experimental group and 30 in the control group.

Data were collected using the Personal Information Form, the Richard-Campbell Sleep Questionnaire (RCSQ), and the Hospital Anxiety and Depression (HAD) Scale.

The patients who underwent open heart surgery and who were in the experimental group were admitted to the ward from the postoperative intensive care unit and the environment was improved for three days based on the improved environment of Watson's HCT, and on the morning of the fourth day in the clinic, the patients were interviewed face to face and the Personal Information Form, RSCQ and HAD Scale were completed. The following improvements were implemented within the scope of environmental improvement:

* Considering the seasonal conditions, the patient room was ensured to have appropriate temperature (18-26 °C) and humidity values (30-60%), and the temperature and humidity were gradually reduced and maintained in the appropriate range by monitoring at 21:00, 22:00, and 23:00 (Days 1, 2, and 3).
* In line with the environmental arrangements, the brightness of the light in the patient room was gradually reduced at 21:00, 22:00, and 23:00 using the Light Meter LM-3000 (Days 1, 2, and 3).

Characteristics of the measuring instrument and application

* The humidity and temperature of the patient room were measured with a Digital-Clock Humidity Meter and Thermometer Device. The Digital-Clock Humidity Meter and Thermometer is a digital thermo-hygrometer that displays indoor temperature and humidity values. The device can stand on the desktop or hang on the wall. The device displays temperature and humidity values, and it also stores the highest and lowest values in its memory. Temperature measurement units can be selected as 0°C or 0°F. The temperature measurement range is -10 to +600, and the accuracy is ± 1 °C. The humidity measurement range of the device with a temperature resolution of 0.1 °C is between 10 and 99%. The humidity sensitivity is ±5%, and the humidity resolution rate is 1%. The device's dimensions are (L) 102 x (W) 21 x (H) 110 mm. It weighed 122 grams.
* The luminous intensity of the light in the patient room was measured with the Light Meter LM-3000 mobile application provided by the researcher. Luminous intensity is the amount of luminous flux per unit area of a surface per unit time. E represents it, lux serves as its unit, and a luxmeter measures it. By definition, we divide the luminous flux of the surface by its area (E = lumen/m2). Light Meter LM-3000 is a mobile application that measures the illuminance of light in lux. Its measurement algorithm offers unrivaled precision to capture the slightest lighting changes, opening up new possibilities in light pollution and health research. Developed by optical scientists and engineers and compatible with five languages, the Light Meter LM-3000 is calibrated using professional Class A equipment for all iPhones and iPads.

The patients in the control group continued to receive standard treatment and care. On the morning of the fourth day after the patients were admitted to the ward from the postoperative intensive care unit, the patients were interviewed face-to-face and the Personal Information Form, RCSQ, and HAD Scale were completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 65 who have undergone open heart surgery and who are conscious and willing to communicate and cooperate.

Exclusion Criteria:

* Patients younger than 18 years and older than 65 years who did not want to participate in the study voluntarily

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Improved sleep quality with optimised environment | The first three days after transfer from intensive care to the ward
  This outcome measure assesses how the improved environment affects postoperative sleep quality with the Richard-Campbell Sleep Questionnaire (RCSQ).
Improvement in anxiety levels with improved environment | The first three days after transfer from intensive care to the ward
  This outcome measure assesses how the improved environment affects postoperative anxiety with the Hospital Anxiety and Depression (HAD) Scale.
Improvement in depression levels with improved environment | The first three days after transfer from intensive care to the ward
  TThis outcome measure assesses how the improved environment affects postoperative depression with the Hospital Anxiety and Depression (HAD) Scale.

CONTACTS AND LOCATIONS:
Overall Officials: HATİCE AZİZOĞLU, Principal Investigator — Study Principal Investigator
Locations (1):
- Yüzüncü Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used to support the findings of this study are available from the corresponding author upon request.

REFERENCES:
- [Result] Nicholson G, Gandra SR, Halbert RJ, Richhariya A, Nordyke RJ. Patient-level costs of major cardiovascular conditions: a review of the international literature. Clinicoecon Outcomes Res. 2016 Sep 21;8:495-506. doi: 10.2147/CEOR.S89331. eCollection 2016. PMID 27703385
- [Result] Yin L, Rong T, Zhang Y, Gao J. The relationship between sleep quality and anxiety and depression among older caregivers of centenarians in China: A cross-sectional study. Geriatr Nurs. 2023 Nov-Dec;54:302-309. doi: 10.1016/j.gerinurse.2023.10.005. Epub 2023 Oct 31. PMID 37918038
- [Result] Frontini R, Rebelo-Goncalves R, Amaro N, Salvador R, Matos R, Morouco P, Antunes R. The Relationship Between Anxiety Levels, Sleep, and Physical Activity During COVID-19 Lockdown: An Exploratory Study. Front Psychol. 2021 Mar 30;12:659599. doi: 10.3389/fpsyg.2021.659599. eCollection 2021. PMID 33859601
- [Result] Demir B, Saritas S. The relationship between anxiety and stress levels with quality of sleep in patients after living donor liver transplantation. Transpl Immunol. 2022 Apr;71:101561. doi: 10.1016/j.trim.2022.101561. Epub 2022 Feb 25. PMID 35219827
- [Result] Nyer M, Farabaugh A, Fehling K, Soskin D, Holt D, Papakostas GI, Pedrelli P, Fava M, Pisoni A, Vitolo O, Mischoulon D. Relationship between sleep disturbance and depression, anxiety, and functioning in college students. Depress Anxiety. 2013 Sep;30(9):873-80. doi: 10.1002/da.22064. Epub 2013 May 16. PMID 23681944
- [Result] Tian Y. A review on factors related to patient comfort experience in hospitals. J Health Popul Nutr. 2023 Nov 8;42(1):125. doi: 10.1186/s41043-023-00465-4. PMID 37941052
- [Result] Wei Q, Lee JH, Park HJ. Novel design of smart sleep-lighting system for improving the sleep environment of children. Technol Health Care. 2019;27(S1):3-13. doi: 10.3233/THC-199002. PMID 31045522
- [Result] Delaney LJ, Currie MJ, Huang HC, Lopez V, Van Haren F. "They can rest at home": an observational study of patients' quality of sleep in an Australian hospital. BMC Health Serv Res. 2018 Jul 5;18(1):524. doi: 10.1186/s12913-018-3201-z. PMID 29976191
- [Result] Yelden K, Duport S, Kempny A, Playford ED. A rehabilitation unit at night: environmental characteristics of patient rooms. Disabil Rehabil. 2015;37(1):91-6. doi: 10.3109/09638288.2014.906662. Epub 2014 Apr 1. PMID 24689441
- [Result] Matsumoto Y, Uchimura N, Ishida T, Morimatsu Y, Mori M, Inoue M, Kushino N, Hoshiko M, Ishitake T. The relationship of sleep complaints risk factors with sleep phase, quality, and quantity in Japanese workers. Sleep Biol Rhythms. 2017;15(4):291-297. doi: 10.1007/s41105-017-0110-1. Epub 2017 Jul 21. PMID 28989323
- [Result] Gimenez MC, Geerdinck LM, Versteylen M, Leffers P, Meekes GJ, Herremans H, de Ruyter B, Bikker JW, Kuijpers PM, Schlangen LJ. Patient room lighting influences on sleep, appraisal and mood in hospitalized people. J Sleep Res. 2017 Apr;26(2):236-246. doi: 10.1111/jsr.12470. Epub 2016 Nov 10. PMID 27862514
- [Result] Falci SG, Marques LS. CONSORT: when and how to use it. Dental Press J Orthod. 2015 May-Jun;20(3):13-5. doi: 10.1590/2176-9451.20.3.013-015.ebo. No abstract available. PMID 26154451
- [Result] Norman V, Rossillo K, Skelton K. Creating Healing Environments Through the Theory of Caring. AORN J. 2016 Nov;104(5):401-409. doi: 10.1016/j.aorn.2016.09.006. PMID 27793250
- [Result] Sarrafzadegan N, Mohammmadifard N. Cardiovascular Disease in Iran in the Last 40 Years: Prevalence, Mortality, Morbidity, Challenges and Strategies for Cardiovascular Prevention. Arch Iran Med. 2019 Apr 1;22(4):204-210. PMID 31126179
- [Derived] Azizoglu H, Gurkan Z, Bozkurt Y, Demir C, Akaltun H. The Effect of an Improved Environment According to Watson's Theory of Human Care on Sleep, Anxiety, and Depression in Patients Undergoing Open Heart Surgery: A Randomized Controlled Trial. Healthcare (Basel). 2025 Jan 18;13(2):183. doi: 10.3390/healthcare13020183. PMID 39857209